CLINICAL TRIAL: NCT05492240
Title: Advancing Rehabilitation Paradigms for Older Adults in Skilled Nursing Facilities
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Colorado, Denver (Other)
Collaborators: Aegis Therapies, Inc. (Unknown); National Institute on Aging (NIA) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 20-3068; R01AG072693 (NIH)
Record Dates: First submitted 2022-07-19; First posted 2022-08-08 (Actual); Last update posted 2026-01-07 (Actual); Status verified 2026-01

CONDITIONS: Aging; Functional Recovery; Skilled Nursing Facility; Medically Complex; Deconditioning
Keywords: Rehabilitation; Older Adults; Physical Therapy; Occupational Therapy; RE-AIM; i-STRONGER; High-intensity Rehabilitation; Implementation Science; Post-Acute Care; Physical Function

STUDY DESIGN:
Who Masked: Participant
Masking Description: Investigators will not be blinded to the arms due to facility/clinician training required for this study design. Study sites [i.e., skilled nursing facilities (SNFs)] will be the unit of randomization. SNF study sites will be made broadly aware of the study initiative during the site recruitment process; however, the site will not be provided with detailed information about the intervention unless randomized to the Intervention arm. As such, clinicians, or rehabilitation care providers, at usual care sites will remain blinded to the intervention for the duration of the study. Clinicians will collect patient-level functional outcomes as part of their standard of care and all patients who are subjects of the intervention will not be aware of the group allocation in the study.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- i-STRONGER (Experimental): The high-intensity rehabilitation intervention, termed i-STRONGER, relies on principles of physiologic overload using an 8-repetition max (8RM) to promote muscle strengthening and emphasizes functional carryover for independence.
  Interventions: Other: i-STRONGER
- Usual Care (Active Comparator): The Usual Care SNFs will continue clinical practice as normal, and sites will not have any overlap of personnel or training with i-STRONGER SNFs.
  Interventions: Other: Usual Care

INTERVENTIONS:
Other: i-STRONGER — An 8RM is the dose necessary for most effective strength gains in community-dwelling older adults, and is equivalent to 80% of a one repetition max, which is the maximal load needed to voluntarily complete one repetition of a given exercise with proper form. Clinicians will tailor the intervention for each activity, so the patient achieves 8 repetitions with failure on the 9th repetition. Failure is the inability to complete a repetition through the full, available range of motion without significant compensation. Further, high-intensity dosing requires continuous, volitional effort from the patient; therefore, incorporation of motivational interviewing strategies across sessions will maximize patient effort and self-efficacy.
  Arms: i-STRONGER
Other: Usual Care — Usual Care SNFs will continue with routine collection and documentation of physical performance outcomes (gait speed, SPPB, Modified Barthel ADL Index) as standard practice. Furthermore, a combination of chart reviews and on-site or remote observation will allow for characterization of usual care components for descriptive comparison. Importantly, the Usual Care SNF including the facility, rehabilitation clinicians, and patients will not have access to i-STRONGER materials.
  Arms: Usual Care

SUMMARY:
This cluster randomized clinical trial seeks to provide large-scale, foundational evidence that high-intensity rehabilitation is effective and can be systematically implemented to improve functional outcomes for patients admitted to skilled nursing facilities following hospitalization. Additionally, this study will generate a descriptive overview of factors that predict implementation success while informing effective implementation strategies for future skilled nursing facilities innovation.

DETAILED DESCRIPTION:
In the U.S., 8.37 million adults over 65 will experience a hospital stay over the next year, which often has serious and long-lasting consequences including profound deterioration in physical function. Following a hospital stay, around 1.35 million patients with deconditioning require rehabilitation in a skilled nursing facility (SNF) each year to address the deleterious musculoskeletal and functional deficits from deconditioning. More than 64% of patients discharge from SNFs at functional levels that predispose them to adverse events, including rehospitalization, failing health, disability, institutionalization, or death. Physical function is a known modifiable predictor of these deleterious events, which can be addressed with rehabilitation. Therefore, more progressive and targeted musculoskeletal rehabilitation strategies that optimize physical function more effectively are needed.

Therefore, the purpose of this study is to determine the effectiveness of a high-intensity rehabilitation approach (also referred to as i-STRONGER) at multiple skilled nursing facilities (SNFs), while evaluating characteristics of successful implementation through a rigorous, pragmatic cluster randomized controlled trial (16 Intervention SNFs vs 16 Usual Care SNFs). The investigators will promote high-intensity rehabilitation delivery to patients in an effort to address poor physical function outcomes. Specifically, the investigators will train rehabilitation clinicians at Intervention sites using distance-based instruction and collect study outcomes via the electronic medical record. Additionally, the investigators will gather quantitative and qualitative data (mixed methods) to evaluate processes, clinician-specific characteristics, and facility-specific contexts of implementation. The study methods seek to maximize successful reach, effectiveness, adoption, implementation, and maintenance (RE-AIM) across Intervention sites. The implementation strategy is informed by the RE-AIM framework and integrated with educational and behavioral theories to facilitate clinical adoption of high-intensity rehabilitation.

ELIGIBILITY:
Rehabilitation staff at enrolled sites will participate in research activities, as indicated by group assignment.

Site Inclusion Criteria:

* Aegis Therapies-contracted skilled nursing facility (SNF)
* Admits approximately 15 patients per month for short term rehabilitation

Patient Inclusion Criteria:

* At least 50 years of age
* Admitted to a SNF from the hospital
* Ambulatory upon SNF admission

Patient Exclusion Criteria:

* Contraindications to high-intensity resistance training, per American College of Sports Medicine Exercise Testing and Prescription
* Lower extremity weight-bearing precautions
* Neurological diagnosis (e.g., Cerebral vascular accident, Multiple Sclerosis, Parkinson's disease)
* Subsequent SNF admission

Ages: 50 Years to 120 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 4383 (Actual)
Dates: Start 2022-07-24 (Actual); Primary Completion 2025-09-16 (Actual); Study Completion 2025-09-16 (Actual)

PRIMARY OUTCOMES:
Change in Gait Speed | From date of admission into the SNF to date of discharge from the SNF, which would be an approximate average of 21 days
  Gait speed will be measured in meters/second using the time it takes to walk a 4-meter path at usual speed using a stopwatch.

SECONDARY OUTCOMES:
Change in Short Physical Performance Battery (SPPB) | From date of admission into the SNF to date of discharge from the SNF, which would be an approximate average of 21 days
  The SPPB is comprised of 3 tasks: a hierarchical standing balance test (side-by-side, semi-tandem, and tandem), a 4-meter usual gait speed, and a 5-time sit-to-stand from a standardized chair. Each subtask is scored (based on time) from 0-4 points and then summarized into a total score of 0-12 points, where 12 points represents the highest performance.
Post-discharge Rehospitalization Rate | From date of discharge from the SNF, assessed up to 30 days
  The proportion of patients eligible for high-intensity rehabilitation who return to the hospital within 30 days of discharge from the SNF.

OTHER OUTCOMES:
Change in Total Score Modified Barthel ADL Index (MBI) | From date of admission into the SNF to date of discharge from the SNF, which would be an approximate average of 21 days
  The Modified Barthel ADL Index assesses the ability to perform basic Activities of Daily Living (ADL) tasks. Total score range is 0-100. Total score is commuted by summing dependence across 10 ADL tasks: chair/bed transfers, ambulation, stair climbing, toilet transfers, bowel control, bladder control, bathing, dressing, personal hygiene (grooming), and feeding. Higher scores indicate increased independence.
RE-AIM Component: Reach | Up to 16 months
  Proportion of patients treated with high-intensity rehabilitation out of all eligible patients.
RE-AIM Component: Adoption | Up to 16 months
  Proportion of clinicians using high-intensity rehabilitation with at least 75% of eligible patients out of all trained clinicians at Intervention sites.
RE-AIM Component: Implementation | Up to 16 months
  Proportion of completed high-intensity rehabilitation elements out of all intervention elements assessed by a fidelity checklist.
RE-AIM Component: Maintenance | Assessed from 16 months up to 22 months
  Proportion of facilities that sufficiently completed high-intensity elements out of all intervention elements assessed by a fidelity checklist.

CONTACTS AND LOCATIONS:
Overall Officials: Jennifer Stevens-Lapsley, PhD, Principal Investigator — University of Colorado, Denver
Locations (2):
- United States (2):
  - University of Colorado Denver, Anschutz Medical Campus, Aurora, Colorado
  - Aegis Therapies, Frisco, Texas

IPD SHARING:
Plan to Share IPD: Yes
The study team guarantees that any and all data collected as part of this project will be released in accordance with standard data sharing policies and procedures to validate research findings if requested. Data will be made available in a timely manner to the broader scientific community, and will be complete, and as accurate as possible. All data released will be de-identified, with no information that could be linked to any study subjects, or participating study practices to ensure the confidentiality of all subjects and practices. If necessary, a data use agreement will be established.
Supporting Information: Study Protocol, SAP, ICF
Time Frame: The data will be available starting 6 months after primary study publication and ending 2 1/2 years after publication.
Access Criteria: Data will be made available upon reasonable written request to the study team. The PI, Dr. Jennifer Stevens-Lapsley will review requests.